CLINICAL TRIAL: NCT00138996
Title: Can the Quality of Cardiopulmonary Resuscitation Improve With Direct Online Feedback From the Defibrillator to the Rescuers on Their Resuscitation Efforts
Brief Title: Quality of Cardiopulmonary Resuscitation Without and With Defibrillator Feedback
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Laerdal Medical (Industry); Ullevaal University Hospital (Other); Health Region East, Norway (Other); Norwegian Air Ambulance Foundation (Other); London Ambulance Service (Other); Stockholm Ambulance Service (Unknown); University of Chicago (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-01139; 2002-OSL-MDD-0009 (DNVeritas)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; resuscitation; quality; feedback; training
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: automated direct feedback on CPR from defibrillator

SUMMARY:
Quality of bystander cardiopulmonary resuscitation (CPR) affect patient survival. Quality of professional CPR on patients has not been studied in detail, but it is regularly reported that the quality when tested on manikins deteriorates dramatically within months after training. Automated direct feedback on CPR quality from manikins brings quality back within a couple of minutes. Similar feedback has been incorporated into a defibrillator which also monitors quality of CPR. We hypothesise that quality of professional clinical CPR improves with such feedback

DETAILED DESCRIPTION:
Defibrillators which monitor quality of CPR via changes in thoracic impedance (for ventilation) and movement of the sternum employing an accelerometer (for chest compressions) will be employed in ambulances in Akershus county (Norway), Stockholm (Sweden) and London (UK). During phase 1 quality of CPR will be monitored without feedback from the defibrillator. During phase 2 the ambulance personnel will receive feedback via the defibrillator. During phase 3 the ambulance personnel will be retrained with particular attention to the quality problems that became apparent in phase 3.

Quality of CPR will be continuously recorded by the defibrillators and the data collected and sent via internet to Laerdal Medical. All other cardiac arrest data including survival will be recorded using standard datasets for cardiac arrest research as developed by a task force with members from the organisations in International Liaison Committee on resuscitation (Utstein guidelines). The data will be annotated and analyzed in detail by researchers at University of Oslo

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest out-of-hospital

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-03; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
fraction of time without CPR
chest compression depth
chest compression frequency
chest compression/decompression duty cycle
ventilation frequency

SECONDARY OUTCOMES:
rate of return of spontaneous circulation

CONTACTS AND LOCATIONS:
Overall Officials: Petter A Steen, Principal Investigator — University of Oslo, Ulleval University Hospital
Locations (3):
- Ulleval University Hospital, Oslo, Norway
- Stockholm Ambulance Service, Stockholm, Sweden
- London Ambulance Service, London, United Kingdom

REFERENCES:
- [Result] Wik L, Kramer-Johansen J, Myklebust H, Sorebo H, Svensson L, Fellows B, Steen PA. Quality of cardiopulmonary resuscitation during out-of-hospital cardiac arrest. JAMA. 2005 Jan 19;293(3):299-304. doi: 10.1001/jama.293.3.299. PMID 15657322
- [Derived] Kramer-Johansen J, Edelson DP, Abella BS, Becker LB, Wik L, Steen PA. Pauses in chest compression and inappropriate shocks: a comparison of manual and semi-automatic defibrillation attempts. Resuscitation. 2007 May;73(2):212-20. doi: 10.1016/j.resuscitation.2006.09.006. Epub 2007 Jan 22. PMID 17241734
- [Derived] Kramer-Johansen J, Myklebust H, Wik L, Fellows B, Svensson L, Sorebo H, Steen PA. Quality of out-of-hospital cardiopulmonary resuscitation with real time automated feedback: a prospective interventional study. Resuscitation. 2006 Dec;71(3):283-92. doi: 10.1016/j.resuscitation.2006.05.011. Epub 2006 Oct 27. PMID 17070980